CLINICAL TRIAL: NCT01695447
Title: Randomised Controlled Trail of Duct-to-mucosa Versus Invagination for Pancreaticojejunostomy After Pancreaticoduodenectomy
Brief Title: Duct-to-mucosa Versus Invagination for Pancreaticojejunostomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: TingBo Liang (Other)
Responsible Party: Sponsor-Investigator, TingBo Liang, The Second Affiliated Hospital, School of Medicine, Zhejiang Universtiy, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZEH-LL-CX-004-02
Record Dates: First submitted 2012-09-20; First posted 2012-09-28 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Pancreatic Neoplasms; Biliary Tract Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- duct-to-mucosa (Experimental): duct-to-mucosa technique is used for pancreaticojejunostomy after pancreaticoduodenectomy
  Interventions: Procedure: duct-to-mucosa; Device: Internal stent
- invagination (Active Comparator): invagination technique is used for pancreaticojejunostomy after pancreaticoduodenectomy
  Interventions: Procedure: invagination; Device: Internal stent

INTERVENTIONS:
Procedure: duct-to-mucosa
  Arms: duct-to-mucosa
Procedure: invagination
  Arms: invagination
Device: Internal stent — Internal stent may be used during pancreaticojejunostomy according to the situation of pancreatic duct and experience of the surgeon.

SUMMARY:
The purpose of this study is to determine whether duct-to-mucosa is better than invagination in pancreaticojejunostomy after pancreaticoduodenectomy. This single-centre, open, randomized controlled trail is conducted following ISGPF criteria for pancreatic fistula (PF). The duration of the study is supposed to start from Jan 5th 2012 and last to Dec 2014, until 100 or more cases are accessible. Patients diagnosed with pancreatic cancer, peri-ampullar carcinoma or other benign or malignant diseases which need to operate pancreaticoduodenectomy will be included. Main outcomes are pancreatic fistula rate, mortality, morbidity, reoperation and hospital stay. The investigators assumption that duct-to-mucosa is better than invagination.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with pancreatic cancer or other diseases which need pancreaticoduodenectomy and pancreaticojejunostomy
* 18 to 80 y/o
* Operation-tolerated
* Informed consent

Exclusion Criteria:

* History of gastrointestinal operation
* Pancreaticoduodenectomy is given up during operation
* Pancreatic duct is difficult to locate
* Patients require to exit from the study anytime

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
pancreatic fistula | From date of operation until the date of dischage or date of death from any cause, whichever came first,, assessed up to 200 days
  The determine of pancreatic fistula follows the International Study Group on Pancreatic Fistulas (ISGPF) criteria.

SECONDARY OUTCOMES:
Mortality | From date of operation until the date of in-hospital death or death within 30 days after operation, whichever came first, assessed up to 200 days
  30-day or in-hospital mortality: death from any cause within 30 days after operation or any in-hospital death are considered concerned with the type of pancreaticojejunostomy
Morbidity | From date of operation until the date of discharge or date of death from any cause, whichever came first, assessed up to 200 days
  any complications after operation will be recorded.
Reoperation | From date of operation until the date of discharge or date of death from any cause, whichever came first, assessed up to 200 days
  Reasons and times of reoperation are recorded. The attending doctor will decided Whether reoperation is needed, according to indications and his experience.
Hospital stay | From date of operation until the date of discharge or date of death from any cause, whichever came first, assessed up to 200 days
  Post-operation hospital stay is assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital, School of Medicine, Zhejiang Universtiy, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Bai X, Zhang Q, Gao S, Lou J, Li G, Zhang Y, Ma T, Zhang Y, Xu Y, Liang T. Duct-to-Mucosa vs Invagination for Pancreaticojejunostomy after Pancreaticoduodenectomy: A Prospective, Randomized Controlled Trial from a Single Surgeon. J Am Coll Surg. 2016 Jan;222(1):10-8. doi: 10.1016/j.jamcollsurg.2015.10.003. Epub 2015 Oct 21. PMID 26577499